CLINICAL TRIAL: NCT00363441
Title: A Randomized Phase II Study of Conventional 3D Radiation (3DCRT) Versus Intensity-Modulated Radiation (IMRT) in Squamous Cell Cancer of the Head and Neck (SCCHN): Pilot Feasibility Study
Brief Title: A Study of Conventional 3D Radiation vs. Intensity-Modulated Radiation in Squamous Cell Cancer of the Head and Neck
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20313
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Head and Neck Neoplasms; Squamous Cell Cancer
Keywords: head and neck neoplasms; squamous cell cancer; intensity modulated radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Procedure: Intensity Modulated Radiotherapy

SUMMARY:
This is a randomized study of conventional 3d radiation versus intensity-modulated radiation in squamous cell cancer of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven squamous cell carcinoma of the head and neck or squamous cell cancer to the neck from an unknown head and neck primary site, stage I-IV disease which is M0, age greater than 18 years, KPS greater than 70, signed study-specific consent

Exclusion Criteria:

* M1; bilateral N3 disease; primary greater than 10cm; salivary gland disease; life expectancy less than 2 years; prior radiotherapy to the head and neck; no signed study-specific consent form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of side effects according to Radiation Therapy Oncology Group
scales and CTCAE version 3.0 for acute and chronic radiation toxicities, local control rates

CONTACTS AND LOCATIONS:
Overall Officials: Harold P Lau, MD, Principal Investigator — Tom Baker Cancer Center